CLINICAL TRIAL: NCT06132607
Title: Evaluating Three-dimensional Lung Reconstructions for Uniportal Thoracoscopic Lung Resections Using Open-source Software
Brief Title: 3D Lung Reconstructions Using Open-source Software for Lung Cancer Surgery
Acronym: 3D-LUNG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Z2022177; METCZ20220105 (Other: METC Z)
Record Dates: First submitted 2023-10-31; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Lung Cancer; Thoracic Surgery, Video-Assisted; Lobectomy; Segmentectomy; Humans; Surgery
Keywords: video-assisted thoracoscopic surgery; lung cancer; three-dimensional reconstruction; three-dimensional simulation; open-source software
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative 3D lung reconstruction (Experimental): Patients who were planned for an anatomical lung resection with preoperative 3D lung reconstruction.
  Interventions: Device: Preoperative 3D lung reconstruction created with open-source software

INTERVENTIONS:
Device: Preoperative 3D lung reconstruction created with open-source software — Preoperative 3D lung reconstruction created with open-source software 3D Slicer
  Other Names: 3D Slicer

SUMMARY:
Preoperative three-dimensional (3D) lung reconstructions can reduce intraoperative blood loss, conversion rate, and operation duration. Commercial products predominantly provide these 3D reconstructions, hence the aim of this study was to assess the usability and performance of preoperative 3D lung reconstructions created with open-source software.

DETAILED DESCRIPTION:
A single-center prospective pilot study is conducted within the thoracic surgery department of the Zuyderland Medical Center, Heerlen, the Netherlands. Patients are recruited during preoperative consultation with the thoracic surgeon. The aim of this study is to include at least 12 patients in this pilot study based on the sample size for pilot studies.

Before the pilot study, the surgeons involved in the study set several requirements for the 3D lung reconstructions. A technical physician, a healthcare professional in the Netherlands who combines knowledge of technology and medicine and is licensed to perform medical interventions, creates three-dimensional lung reconstructions using open-source 3D Slicer software that fulfills these aforementioned requirements and uses the available preoperative diagnostic late arterial phase contrast-enhanced CT scans.

Three thoracic surgeons (with at least five years of uniportal VATS experience) and one surgical resident in thoracic surgery assess these 3D lung reconstructions for preoperative planning of uniportal VATS anatomical resections and compare the outcome measures based on the 3D lung reconstructions with the 2D CT scan and intraoperative findings.

Patient characteristics, including age, sex, Eastern Cooperative Oncology Group (ECOG) performance status, body mass index, American Society of Anesthesiologists classification, forced expiratory volume in 1s (FEV1), diffusion capacity of the lung for carbon monoxide by the single-breath technique (DLCO-SB), intoxications, clinical Tumor Nodule Metastasis (TNM) classification 8th edition, previous thoracic surgery, and comorbidities are extracted from patient records. The following perioperative and postoperative data are collected: surgical approach, planned lung resection, performed lung resection, surgery duration, conversion, blood loss, surgery difficulty, the radicality of resection, pathological TNM classification 8th edition, tumor size, final pathology, drain duration, length of hospital stay, and complications within 30 days of surgery. The difficulty of the surgical procedure will be assessed by the thoracic surgeon and rated on a 5-point Likert scale from 1 (very easy) to 5 (very difficult). Length of hospital stay is defined as the number of days between the first day after surgery and the day the patient was clinically discharged.

Descriptive statistical analyses are performed in IBM SPSS Statistics v28 (MacOS, Armonk, New York, United States). Missing data will be reported as such.

ELIGIBILITY:
Inclusion Criteria:

Patients with suspected or biopsy-proven lung cancer scheduled for video-assisted thoracoscopy surgery for lobectomy or segmentectomy

Exclusion Criteria:

* Computed Tomography scan contained motion artifacts
* Surgery was canceled
* Planned surgery changed intraoperatively to another procedure
* Patients who did not provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
System Usability Score | Single-point evaluation after surgery (at day 0)
  System Usability Score Questionnaire. This questionnaire includes 10 statements rated from 1 (strongly disagree) to 5 (strongly agree). The even-numbered questions contributed to the scale position 5 minus the scale position, while the odd-numbered questions contributed to the scale position minus 1. The final score was calculated by the sum of the even and uneven-numbered questions, multiplied by 2.5. The minimum system usability score is 0 and the maximum is 100. A system usability score above 68 is considered above average.

SECONDARY OUTCOMES:
Segmental lung nodule location | Baseline and during surgery (at day 0)
  The performance of the 3D lung reconstructions is evaluated based on the anatomical validity of the 3D lung reconstructions compared to the two-dimensional (2D) CT scan and intraoperative findings. Before surgery, a number of anatomical components of the 3D lung reconstructions are assessed. During surgery, the anatomical validity of these anatomical components is verified. One of the anatomical components includes the segmental location of the lung nodule.
Number of arteries to target lobe or segment | Baseline and during surgery (at day 0)
  The performance of the 3D lung reconstructions is evaluated based on the anatomical validity of the 3D lung reconstructions compared to the two-dimensional (2D) CT scan and intraoperative findings. Before surgery, a number of anatomical components of the 3D lung reconstructions are assessed. During surgery, the anatomical validity of these anatomical components is verified. One of the anatomical components includes the number of arteries towards the target lobe or segment.
Anatomical variations | Baseline and during surgery (at day 0)
  The performance of the 3D lung reconstructions is evaluated based on the anatomical validity of the 3D lung reconstructions compared to the two-dimensional (2D) CT scan and intraoperative findings. Before surgery, a number of anatomical components of the 3D lung reconstructions are assessed. During surgery, the anatomical validity of these anatomical components is verified. One of the anatomical components includes the presence of (a) anatomical variation(s).
Potential change of surgery or surgical plan | Single-point evaluation after surgery (at day 0)
  As another part of the evaluation of the performance, the potential impact of the 3D lung reconstructions on the surgical plan was also considered. Therefore, the surgeon was asked after surgery if the 3D lung reconstruction would have resulted in a preoperative change in surgical approach.
Intraoperative use of 3D lung reconstruction | Single-point evaluation after surgery (at day 0)
  As final part of the evaluation of the performance, the potential value during surgery of the 3D lung reconstructions was also considered. Therefore, the surgeon was asked after surgery whether they would like to have used the 3D lung reconstruction during surgery via a tablet for example.

CONTACTS AND LOCATIONS:
Overall Officials: Erik de Loos, PhD, Principal Investigator — Department of Surgery, Zuyderland Medical Center, Heerlen, the Netherlands
Locations (1):
- Zuyderland Medical Center, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author, ER de Loos, upon reasonable request.

REFERENCES:
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharm Stat 2005;4:287-91.
- [Background] Lewis JR, Sauro J. Item benchmarks for the system usability scale. J Usability Stud 2018;13.
- [Background] Brooke J. SUS: a 'quick and dirty' usability. Usability Eval Ind 1996;189:189-94.
- [Derived] Laven IEWG, Oosterhoff VPS, Franssen AJPM, van Roozendaal LM, Hulsewe KWE, Vissers YLJ, de Loos ER. Evaluating three-dimensional lung reconstructions for thoracoscopic lung resections using open-source software: a pilot study. Transl Lung Cancer Res. 2024 Jul 30;13(7):1595-1608. doi: 10.21037/tlcr-24-134. Epub 2024 Jul 16. PMID 39118878